CLINICAL TRIAL: NCT05011266
Title: Efficacy of Buprenorphine and XR-Naltrexone Combination for Relapse Prevention in Opioid Use Disorder
Acronym: COMBO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB #8171; U01DA046430 (NIH)
Record Dates: First submitted 2021-08-16; First posted 2021-08-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder
Keywords: opioid use disorder; treatment; buprenorphine; extended release naltrexone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: parallel arm, double-blind, placebo-controlled buprenorphine compared to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buprenorphine-naloxone (Experimental): Buprenorphine/naloxone 5.7 mg /1.4 mg/day sub-lingual tablets
  Interventions: Drug: Buprenorphine/naloxone
- Placebo (Placebo Comparator): placebo sub-lingual tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine/naloxone — 5.7 mg buprenorphine/1.4 mg naloxone sub-lingual daily
  Other Names: Zubsolv
  Arms: Buprenorphine-naloxone
Drug: Placebo — placebo sub-lingual tablet daily
  Other Names: PBO
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of a new pharmacological approach to increase efficacy of treatment with extended release naltrexone (XR-naltrexone) for individuals with opioid use disorder by combining it with buprenorphine-naloxone. This is a two arm, double-blind, placebo-controlled study to examine whether addition of buprenorphine-naloxone will improve treatment retention, reduce opioid craving, and improve mood over 24 weeks of treatment with extended release naltrexone (XR-naltrexone) administered every four weeks for a total of 6 injections.

The NYSPI site, which provides study oversight (no direct participant involvement) is currently paused and has been paused since an institutional pause on human subjects research began in June, 2023. The U.S. Department of Health and Human Services (HHS) Office of Human Research Protections (OHRP) issued an FWA restriction on NYSPI research that also included a pause of human subjects research as of June 23, 2023.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of a new pharmacological approach to increase efficacy of treatment with extended release naltrexone (XR-naltrexone) for individuals with opioid use disorder by combining it with buprenorphine-naloxone. Adding buprenorphine-naloxone after the patient initiated XR-naltrexone will not produce mu opioid agonist effect but kappa antagonist effects of buprenorphine may provide additional relief of protracted withdrawal, craving, and mood disturbances persisting in patients treated with XR-naltrexone and possibly contributing to premature treatment discontinuation and relapse. This is a parallel arm, double-blind, placebo-controlled study to examine whether addition of buprenorphine will improve treatment retention, reduce opioid craving, and improve mood over 24 weeks of treatment with XR-naltrexone administered every four weeks. Individuals with Opioid Use Disorder (OUD) and beginning treatment with XR-naltrexone for maintenance treatment will be randomized to treatment with adjunctive buprenorphine-naloxone or placebo with 5 additional doses of XR-naltrexone, given every four weeks, and weekly medication management. The study will provide detoxification and a first XR-Naltrexone injection if a participant consents before the first XR-naltrexone injection. In all participants randomization will occur after first XR-NTX injection. Buprenorphine-naloxone (sub-lingual (SL), 4/1 mg/day) or placebo will be started after a first XR-naltrexone dose and tapered off at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65 (inclusive) interested in antagonist-based relapse prevention treatment
* Meets current DSM-5 criteria for current opioid use disorder of at least six months duration supported by urine toxicology positive for opioids OR positive naloxone challenge (defined by 3-point increase in COWS) if seeking detoxification and XR-NTX induction OR confirmed recent detoxification treatment for opioids.
* In otherwise good health based on complete medical history, physical examination, vital signs measurement, ECG, and laboratory tests (hematology, blood chemistry, urinalysis) with no clinically significant abnormalities
* Participants who completed detoxification and received XR-NTX are eligible for the study. Participants may be enrolled up to 2 weeks following an initial XR-NTX injection given in any outside research or community-based treatment setting (inpatient, outpatient residential).
* Seeking treatment for opioid use disorder, willing to accept treatment with XR-NTX and, in the judgment of the treating physician, is a good candidate for naltrexone-based treatment.
* Voluntarily seeking treatment for opioid use disorder.
* Able to give written informed consent to participate in the study and showing a thorough understanding of the difference between agonist and antagonist-based treatment.

Exclusion Criteria:

* Methadone maintenance within 2 weeks of XR-NTX induction or any use of methadone in the week prior to XR-NTX induction
* Maintenance on buprenorphine or frequent buprenorphine use in the week prior to XR-NTX induction (must be using no more than 8 mg of buprenorphine per day for no more than 3 days per week). If consenting after initial XR-NTX injection, any use of buprenorphine since XR-NTX induction is exclusionary.
* Serious medical, psychiatric or substance use disorder that, in the opinion of the study physician, would make a detoxification and naltrexone initiation, or maintenance treatment with XR-NTX in combination with buprenorphine, hazardous (relative contraindications) or requires a different level of care. Examples include:

  1. Disabling or terminal medical illness (e.g., uncompensated heart failure, severe acute hepatitis, cirrhosis or end-stage liver disease) as assessed by medical history and/or review of systems.
  2. Severe, untreated or inadequately treated mental disorder (e.g., active psychosis, uncontrolled manic-depressive illness) as assessed by history and/or clinical interview.
  3. Current severe alcohol, benzodiazepine, or other depressant or sedative hypnotic use likely to require a complicated medical detoxification (routine alcohol and sedative detoxifications may be included).
  4. Suicidal or homicidal
* AST/ALT > 3x normal limit
* Pregnancy, lactation, or a plan of becoming pregnant. Women need to have negative blood pregnancy test at screening and agree to practice dual contraceptives.
* Physiological dependence on alcohol or sedative-hypnotics with impending withdrawal. Other substance use diagnoses are not exclusionary.
* History of allergic or adverse reaction to buprenorphine, naltrexone, naloxone, clonidine, or clonazepam.
* Painful medical condition that requires ongoing opioid analgesia or anticipated surgery necessitating opioid medications.
* Individuals above 60 with possible early cognitive decline or other neurodegenerative conditions as evidenced by a score of less than 25 on a Mini Mental Status Exam screen.
* Participants who had 30 or more opioid-free days prior to randomization will not be eligible.
* Participants more than 2 weeks following an initial XR-NTX injection (given in any outside research or community-based treatment setting, for example inpatient, outpatient residential).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants receiving XR-naltrexone injections | 20 weeks
  Proportion of patients successfully retained to receive six consecutive XR-naltrexone injection.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, MD, Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - Avery Road Treatment Center (ARTC), Rockville, Maryland
  - Stars/Nyspi, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published in this report (after de-identification) (text, tables, figures)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning twelve months and ending 5 years after article publication
Access Criteria: to researcher who provides a methodologically sound proposal to achieve aims in approved proposal
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086